CLINICAL TRIAL: NCT01752166
Title: Prospective Collection and Testing of Un-Spiked and Candida-Spiked Fresh Whole Blood Specimens From Patients Who Have Been Referred For a Diagnostic Blood Culture
Brief Title: Detecting Infections Rapidly and Easily for Candidemia Trial - Part 2 (direcT2 Study)
Acronym: direcT2
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00031
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Candidemia
Keywords: Candida; Candidemia; Blood culture; Diagnostics
MeSH Terms: conditions — Candidemia; Torulopsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood culture: Subjects have had a blood culture ordered, per routine standard of care

SUMMARY:
The purpose of this study is to validate clinical performance (i.e. estimated sensitivity and specificity) of the T2 Candida test on the T2 DX Instrument compared to blood culture results and/or known Candida positive status of prospectively collected and contrived (i.e. Candida-spiked) clinical specimens.

DETAILED DESCRIPTION:
This study will prospectively collect and analyze whole blood T2 clinical research specimens and concomitant blood culture specimens from patients who have been referred for a blood culture per routine standard of care. Additional analysis of blinded, contrived (i.e. Candida spiked and un-spiked whole blood) specimens will be completed by study sites to augment the analysis of Candida positive blood specimens prospectively obtained from the study population.

The clinical performance of the T2 Candida test on the T2 Dx Instrument will be evaluated by calculating the:

* Estimated clinical specificity of the T2Candida test results compared to Candida negative blood culture results in prospectively collected specimens, and the
* Estimated sensitivity of the T2 Candida test results compared to the known Candida positive status or Candida positive blood culture status of contrived specimens that have been spiked at clinically relevant concentrations of the target organisms and, where detected, to Candida positive blood culture results in prospectively collected clinical specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's authorized representative must be able to understand, read and sign the study specific informed consent form after the nature of the study has been fully explained to them.
2. Subject has had a blood culture ordered, per routine standard of care.
3. Subject is between 18-95 years of age

Exclusion Criteria:

1. Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study.
2. Subject has had previous specimens tested by the T2Candida assay with valid results.
3. Subject has had an anti-fungal drug administered through the same port or central line as is used to collect the clinical research specimens.
4. Treatment of subject with any novel drug compound within 30 days prior to the collection of T2 blood specimens.
5. T2 clinical specimen, Tube A contains <3ml of blood.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have had a blood culture ordered, per routine standard of care
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Specificity | Up to 19 hours post blood collection
  Estimated specificity of the T2Candida test will be examined by comparing T2Candida test results from prospectively collected T2 clinical specimens to blood culture results from specimens that are culture negative for Candida and which have been collected at the same time and from the same anatomical location as the T2 specimens.
Sensitivity | Up to 19 hours post blood collection
  Estimated sensitivity of the T2Candida test will be examined by comparing T2Candida test results to the known Candida positive status or Candida positive blood culture status of contrived specimens that have been spiked at clinically relevant concentrations of the target organisms and, where detected, to blood culture results from specimens that are culture positive for Candida and which have been collected at the same time and from the same anatomical location as the T2 specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pappas, MD, Principal Investigator — University of Alabama at Birmingham
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgia Regents University, Augusta, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Houston College of Pharmacy, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas

REFERENCES:
- [Derived] Mylonakis E, Clancy CJ, Ostrosky-Zeichner L, Garey KW, Alangaden GJ, Vazquez JA, Groeger JS, Judson MA, Vinagre YM, Heard SO, Zervou FN, Zacharioudakis IM, Kontoyiannis DP, Pappas PG. T2 magnetic resonance assay for the rapid diagnosis of candidemia in whole blood: a clinical trial. Clin Infect Dis. 2015 Mar 15;60(6):892-9. doi: 10.1093/cid/ciu959. Epub 2015 Jan 12. PMID 25586686